CLINICAL TRIAL: NCT03460808
Title: The Combination of Atorvastatin, Acetylcysteine and Danazol as the Treatment of Steroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-hui Zhang, Professor, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z171100001017084
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Immune Thrombocytopenia
Keywords: steroid-resistant; refractory; Atorvastatin; Acetylcysteine; Danazol
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Atorvastatin; Acetylcysteine; Danazol; deanol aceglutamate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- atorvastatin, acetylcysteine & danazol (Experimental): atorvastatin 20mg qd po plus acetylcysteine 400mg tid po plus danazol 200mg bid po for 12 weeks
  Interventions: Drug: atorvastatin; Drug: Acetylcysteine; Drug: Danazol

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin was used in combination with acetylcysteine and danazol.
Drug: Acetylcysteine — Acetylcysteine was used in combination with atorvastatin and danazol.
Drug: Danazol — Danazol was used in combination with atorvastatin and acetylcysteine or as the monotherapy
  Other Names: Danocrine; Cleregil; Danol

SUMMARY:
Single-arm, open-lable, multicentre study to compare the efficacy and safety of atorvastatin, acetylcysteine plus danazol with danazol monotherapy in patients with corticosteroidresistant/relapsed ITP.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is a severe bleeding disorder. Approximately 2/3 of patients achieve remission from first-line therapies. However, the underlying mechanism of corticosteroid-resistant or relapsed ITP is not well understood; thus, treatment remains a great challenge. Atorvastatin was shown to enhance bone marrow endothelial cell function and N-acetylcysteine (NAC) was shown to inhibit PLT binding to endothelial cell.

A multicentre prospective study was performed in non-splenectomized ITP patients who were either resistant to a standard dose of corticosteroids or had relapsed. Patients were randomized to atorvastatin, acetylcysteine plus danazol with danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study, in order to compare the efficacy and safety of atorvastatin, acetylcysteine plus danazol with danazol monotherapy in patients with corticosteroid-resistant/relapsed ITP.

ELIGIBILITY:
Inclusion Criteria:

* ITP confirmed by excluding other supervened causes of thrombocytopenia;
* Platelet count of less than 30×10^9/L at enrollment;
* Patients who did not achieve a sustained response to treatment with full dose corticosteroids for a minimum duration of 4 weeks or who relapsed during steroid-tapering or after its discontinuation;
* ECOG<2.
* EPCs in bone marrow less than 0.02%

Exclusion Criteria:

* Secondary immune thrombocytopenia (e.g., patients with HIV, HCV, Helicobacter pylori infection or patients with systemic lupus erythematosus)
* congestive heart failure
* severe arrhythmia
* nursing or pregnant women
* aspartate aminotransferase and alanine transaminase levels ≥ 3× the upper limit of the normal threshold criteria
* creatinine or serum bilirubin levels each 1.5 times or more than the normal range
* active or previous malignancy
* Unable to do blood routine test for the sake of time, distance, economic issues or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
the sustained platelet response at the 6-month follow-up | From the start of study treatment (Day 1) up to the end of Month 6
  The number of participants (responders) with platelet count >=30x10^9/L and at least a 2-fold increase in the baseline count (PR) or a platelet count >=100x10^9/L (CR) and the absence of bleeding, without rescue medication at 6-month follow-up.

SECONDARY OUTCOMES:
overall response | From the start of study treatment (Day 1) up to the end of Month 6
  The number of participants with platelet count >=30×10^9/L at least once and at least a doubling of the baseline platelet count without the administration of any other platelet increasing therapy.
time to response | From the start of study treatment (Day 1) up to the end of Year 2
  Time to response was defined as the time from starting treatment to the time to achieve the response.
duration of response | From the start of study treatment (Day 1) up to the end of Year 2
  Duration of response was measured from the achievement of response to the loss of response.
incidence of treatment-emergent adverse events | From the start of study treatment (Day 1) up to the end of Year 2
  All patients were assessed for treatment-emergent adverse events every week during the first 8 weeks of treatment, and at 2-week intervals thereafter. Adverse events were scaled according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China